CLINICAL TRIAL: NCT00664404
Title: Pharmacogenetics, Emotional Reactivity and Smoking Cessation: Genetic Differences in Limbic Activation Associated With Nicotine Withdrawal
Brief Title: Genetic Differences in Limbic Activation Associated With Nicotine Withdrawal
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2005-0829
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Smoking
Keywords: Smoking; Smoking Cessation; Nicotine Withdrawal; Nicotine Dependence; Neuroregulatory Effects; Magnetic Resonance Imaging; MRI
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- fMRI (Other): Functional Magnetic Resonance Imaging (fMRI)
  Interventions: Other: Functional Magnetic Resonance Imaging (fMRI)

INTERVENTIONS:
Other: Functional Magnetic Resonance Imaging (fMRI) — Functional Magnetic Resonance Imaging (fMRI)of the Brain, one session while smoking, and one session while abstinent from smoking (not smoking).

SUMMARY:
Objectives:

* To evaluate neural correlates associated with emotional processing during nicotine withdrawal preferentially involving the amygdala and associated areas within the corticolimbic and mesolimbic circuitry. We hypothesize that relative to a pre-quit baseline, post-quit nicotine withdrawal will result in increased activity to negative emotional cues, in contrast to other cues, in one or more areas of interest, and particularly in the right cerebral hemisphere.
* To determine if bupropion and varenicline moderate patterns of brain activation during post-quit nicotine withdrawal. We hypothesize that relative to placebo, bupropion and varenicline will attenuate the effects of post-quit nicotine withdrawal on emotional processing, reducing activation to negative emotional cues, relative to other cues, in one or more areas of interest, and particularly in the right cerebral hemisphere.
* To determine if genotype (DRD2 TaqA2 allele and the ins variant of the -141C ins/del DRD2) moderates patterns of brain activation during post-quit nicotine withdrawal.

DETAILED DESCRIPTION:
Before you begin participation in this study, you will be asked to provide the names and addresses of 3 contacts (family member/friends) who will know your current contact information. This is so study researchers can stay in contact with you throughout the study. This is in case study researchers may need to reach you in order to reschedule your appointment time. You will also be asked to sign a letter giving your contacts permission to provide your contact information to the study staff.

If the staff is not able to reach you, they may try to locate you through telephone directory assistance or the internet. If the study staff is still unable to locate you, they may use a locator service, such as Transunion or the National Change of Address (NCOA) database, which is maintained by the United States Postal Service.

If you agree to take part in this study, you will be asked to come to the Behavioral Science Research Clinic at M. D. Anderson for up to 2 laboratory sessions. One session will be while you are smoking, and one session will be while you are abstinent from smoking (not smoking).

At each of these sessions, you will have functional magnetic resonance imaging (fMRI) of your brain while you are looking at slides. fMRI involves a scanner that uses a large magnet, instead of x-rays, to take pictures of the inside of your body. The slides will include pictures of people, nature scenes, artwork, victims of car crashes, medical procedures (such as open surgery or autopsy), and nude people. You will be shown examples of these slides before having the fMRI, and you will be given the opportunity to withdraw from this study at that time. If you choose to continue on this study, you will have an fMRI taken of your brain. This will involve being passed into a narrow tube-shaped scanner that is open at both ends. During the fMRI, your brain electrical activity will be monitored. The total time for each lab session will last about 1.5 hours.

You should not drink more than 2 cups of coffee or other caffeine drinks at least 2 1/2 hours before each session. This is because caffeine may affect brain functioning. Before one or both of your sessions, you may be asked to not smoke from bedtime on the day before the session until after the session on the next day. Before one or both of your sessions, you may be asked to smoke as you would regularly. Additionally, you may be asked to smoke during one or both of your laboratory sessions.

At each lab session, you will be asked to blow air through a carbon monoxide (CO) measuring device. CO is a gas that is found (in higher levels) in the bodies of cigarette smokers. You will also be asked questions about your smoking habits; your health and medical condition; and about any medications you are taking. You will also be asked to complete some questionnaires that will ask about your mood and feelings. You may be asked to complete these questionnaires before, during, or after the fMRI.

At the end of this study, you will be able to ask questions about the results of this study and about procedures you have experienced during this study.

Your participation in this part of the study will last about 2 weeks. It will end after your last lab session. You will still be considered a participant in the main study (Protocol 2003-1024) and may have additional visits, questionnaires, and other activities to complete.

This is an investigational study. Up to 72 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be a participant in 'Pharmacogenetics, Emotional Reactivity & Smoking' (protocol 2003-1024).
2. Both parents must be of European descent. The sample will be limited to individuals of European descent because the majority of the published work on the genes of interest has been limited to this racial group. This has been done mostly to prevent population stratification in genetic studies, since allele frequency differences often exist among groups with differing continents of origin.
3. Right handed. The sample is limited to right handed individuals since we will analyze our neuroimaging data for lateralization effects and inclusion of participants of mixed handedness could confound the results.
4. Age: 18 years or older

Exclusion Criteria:

1. Contraindications for MR imaging procedures (e.g., subjects with certain types of implanted medical devices, such as pacemakers, neurostimulators, etc., or subjects who are claustrophobic).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-04; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Stimulus type (positive, negative, neutral, cigarette) by group (Bupropion/ Varenicline/Placebo) | Pre-quit to 1-2 days post-quit

CONTACTS AND LOCATIONS:
Overall Officials: Paul Cinciripini, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org